CLINICAL TRIAL: NCT00317473
Title: Double-blind,Randomized,Controlled,Dose Escalation Phase 1 Trial in 12-47 Month Old Children in Western Kenya to Evaluate the Safety and Immunogenicity of WRAIR's MSP-1(FMP1) Malaria Vaccine Adjuvanted in GSK's AS02A Versus Rabies Vaccine.
Brief Title: Phase 1 Trial of a Malaria Vaccine in Young Kenyan Children
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Collaborators: Kenya Medical Research Institute (Other); Walter Reed Army Institute of Research (WRAIR) (U.S. Federal Agency); The PATH Malaria Vaccine Initiative (MVI) (Other); United States Agency for International Development (USAID) (U.S. Federal Agency); GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: WRAIR 1030; HSRRB Log No. A-12094 (Other: IRB); KEMRI SSC No. 761 (Other: Ethics Committee); HSPC No. HS171 (Other)
Record Dates: First submitted 2006-04-20; First posted 2006-04-24 (Estimated); Results first posted 2017-10-02 (Actual); Last update posted 2017-10-02 (Actual); Status verified 2017-05

CONDITIONS: Plasmodium Falciparum Malaria
Keywords: Vaccine; Phase 1; Plasmodium falciparum; Malaria; Merozoite surface protein-1; MSP-1; Falciparum malaria protein 1; FMP-1; AS02A
MeSH Terms: conditions — Malaria, Falciparum; Malaria

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- FMP1/AS02A Malaria vaccine 10ug (Experimental): Subject vaccinated with 10 ug of FMP1/AS02A on days 0, 29 and 57
  Interventions: Biological: FMP1/AS02A Malaria vaccine
- FMP1/AS02A Malaria vaccine 25 ug (Experimental): Subject vaccinated with 25 ug of FMP1/AS02A on days 14, 42, and 70
  Interventions: Biological: FMP1/AS02A Malaria vaccine
- FMP1/AS02A Malaria vaccine 50 ug (Experimental): Subject vaccinated with 50 ug of FMP1/AS02A on days 28, 56 and 84
  Interventions: Biological: FMP1/AS02A Malaria vaccine
- Imovax Rabies Vaccine (Active Comparator): Subject vaccinated with Imovax Rabies Vaccine on corresponding FMP1/AS021 vaccination days
  Interventions: Biological: Imovax Rabies vaccine

INTERVENTIONS:
Biological: FMP1/AS02A Malaria vaccine — Subjects vaccinated with FMP1/AS02 vaccine
  Arms: FMP1/AS02A Malaria vaccine 10ug; FMP1/AS02A Malaria vaccine 25 ug; FMP1/AS02A Malaria vaccine 50 ug
Biological: Imovax Rabies vaccine — Subjects vaccinated on corresponding FMP1/AS02A vaccination days
  Arms: Imovax Rabies Vaccine

SUMMARY:
To assess the safety and reactogenicity of the FMP-1/AS02A malaria vaccine in malaria-exposed children living in western Kenya and aged 12-47 months

DETAILED DESCRIPTION:
Study consists of 3 cohorts (12 to 23 months, 24 to 35 months, and 36 to 47 months). Within each cohort subjects were randomized in a 2:1 ration to receive one of three dose levels of FMP1/AS02A (Cohort A, 10 ug; Cohort B, 25 ug; Cohort C, 50 ug) or Imovax Rabies vaccine. Immunization was staggered among dose cohorts; subjects in Cohort B received their first immunization only after the Local Medical Monitor and Data Safety Monitoring Board reviewed Cohort A safety data for the eight-day follow-up period following their first immunization. The same procedure was followed for the immunization of Cohort C. This will be conducted in western Kenya a the Walter Reed Project Lumbewa Clinic.

ELIGIBILITY:
Inclusion Criteria:

* A healthy male or female child, 12 to 47 months of age at the time of screening.
* Written informed consent obtained from at least one parent before study start.
* Available to participate for the duration of the study (12 months).

Exclusion Criteria:

* Acute disease at the time of entry into the study
* Axillary temperature of 37.5 degrees C
* Respiratory rate 50
* Serum ALT 45 IU/l (i.e., > 1.5 X ULN)
* Decreased renal function: serum creatinine levels > 92.2 mM/l (> 1.1 mg/dl).
* Significant anemia (Hgb <8 gm/dL).
* Thrombocytopenia (Platelets < 100,000 per mm3)
* Impaired immunity: (Absolute lymphocyte count [ALC] for 1 year olds < 4.0 x 103/mm3; for 2 year olds < 3.0 x 103/mm3; for 3 year olds < 2.0 103/mm3.
* History of homozygous sickle cell disease (SS).
* Malnutrition (Z score; Malnutrition = Weight for height < - 3 z scores)
* Blood transfusion or use of blood-based product in previous 6 months.
* Prior receipt of a rabies vaccine or an investigational malaria vaccine.
* Use of any investigational drug or vaccine other than the study vaccine within 30 days preceding the first dose of study vaccine, or planned use up to 30 days after the third dose.
* Administration of chronic (defined as more than 14 days) immunosuppressants or other immune-modifying drugs within six months of vaccination. (For cortico-steroids, this will mean prednisone, or equivalent, greater than or equal to 0.5 mg/kg/day. Inhaled and topical steroids are allowed).
* Administration or anticipated administration of a vaccine not foreseen by the study protocol within 30 days of the first dose of vaccine(s) with the exception of tetanus toxoid.
* Previous vaccination with a vaccine containing MPL or QS21 (e.g., RTS,S).
* Any confirmed or suspected immunosuppressive or immunodeficient condition, including human immunodeficiency virus (HIV) infection. (No HIV testing will be undertaken as part of this study.)
* History of allergic reactions or anaphylaxis to immunizations or to any vaccine components.
* History of surgical splenectomy.
* Administration of immunoglobulins or any blood products within the 3 months preceding the first dose of study vaccine or planned administration during the study period.
* Simultaneous participation in any other clinical trial.
* Acute or chronic cardiovascular, pulmonary, hepatic or renal condition, which in the opinion of the PI may increase the risk to the subject from participating in the study.
* Any other condition or circumstance that in the opinion of the investigator may pose a threat to the subject.

Ages: 12 Months to 47 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 135 (Actual)
Dates: Start 2003-06; Primary Completion 2004-07 (Actual); Study Completion 2005-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark R. Withers, M.D., MPH, Principal Investigator — USAMRU-K
Locations (1):
- Walter Reed Project Kombewa Clinic, Kombewa, Nyanza Province, Kenya

IPD SHARING:
Plan to Share IPD: Yes
Kenya Medical Research Institute; WRAIR; The Path Malaria Vaccine Initiative; United States Agency for International Development; GlaxoSmith Kline

REFERENCES:
- [Background] Pichyangkul S, Gettayacamin M, Miller RS, Lyon JA, Angov E, Tongtawe P, Ruble DL, Heppner DG Jr, Kester KE, Ballou WR, Diggs CL, Voss G, Cohen JD, Walsh DS. Pre-clinical evaluation of the malaria vaccine candidate P. falciparum MSP1(42) formulated with novel adjuvants or with alum. Vaccine. 2004 Sep 28;22(29-30):3831-40. doi: 10.1016/j.vaccine.2004.07.023. PMID 15364429
- [Background] Ockenhouse CF, Angov E, Kester KE, Diggs C, Soisson L, Cummings JF, Stewart AV, Palmer DR, Mahajan B, Krzych U, Tornieporth N, Delchambre M, Vanhandenhove M, Ofori-Anyinam O, Cohen J, Lyon JA, Heppner DG; MSP-1 Working Group. Phase I safety and immunogenicity trial of FMP1/AS02A, a Plasmodium falciparum MSP-1 asexual blood stage vaccine. Vaccine. 2006 Apr 5;24(15):3009-17. doi: 10.1016/j.vaccine.2005.11.028. Epub 2005 Nov 28. PMID 16356603
- [Background] Stoute JA, Gombe J, Withers MR, Siangla J, McKinney D, Onyango M, Cummings JF, Milman J, Tucker K, Soisson L, Stewart VA, Lyon JA, Angov E, Leach A, Cohen J, Kester KE, Ockenhouse CF, Holland CA, Diggs CL, Wittes J, Heppner DG Jr; MSP-1 Malaria Vaccine Working Group. Phase 1 randomized double-blind safety and immunogenicity trial of Plasmodium falciparum malaria merozoite surface protein FMP1 vaccine, adjuvanted with AS02A, in adults in western Kenya. Vaccine. 2007 Jan 2;25(1):176-84. doi: 10.1016/j.vaccine.2005.11.037. Epub 2005 Dec 7. PMID 16388879
- [Result] Angov E, Aufiero BM, Turgeon AM, Van Handenhove M, Ockenhouse CF, Kester KE, Walsh DS, McBride JS, Dubois MC, Cohen J, Haynes JD, Eckels KH, Heppner DG, Ballou WR, Diggs CL, Lyon JA. Development and pre-clinical analysis of a Plasmodium falciparum Merozoite Surface Protein-1(42) malaria vaccine. Mol Biochem Parasitol. 2003 May;128(2):195-204. doi: 10.1016/s0166-6851(03)00077-x. PMID 12742586

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subject were randomized in a 2:1 ratio between the FMP1/AS02A and Imovax vaccine groups.
Groups:
- FMP1/AS02A Malaria Vaccine 10ug (Cohort A): Subject vaccinated with 10 ug of FMP1/AS02A on days 0, 29 and 57
  FMP1/AS02A Malaria vaccine: Subjects vaccinated with FMP1/AS02 vaccine
- Imovax (Cohort A); Imovax (Cohort B): Subject vaccinated with Imovax Rabies Vaccine on corresponding FMP1/AS021 vaccination days
- FMP1/AS02A Malaria Vaccine 25 ug (Cohort B): Subject vaccinated with 25 ug of FMP1/AS02A on days 14, 42, and 70
  FMP1/AS02A Malaria vaccine: Subjects vaccinated with FMP1/AS02 vaccine
- FMP1/AS02A Malaria Vaccine 50 ug (Cohort C): Subject vaccinated with 50 ug of FMP1/AS02A on days 28, 56 and 84
  FMP1/AS02A Malaria vaccine: Subjects vaccinated with FMP1/AS02 vaccine
- Imovax (Cohort C): Subject vaccinated with Imovax Rabies Vaccine on corresponding FMP1/AS021 vaccination days
  Imovax Rabies vaccine: Subjects vaccinated on corresponding FMP1/AS02A vaccination days
Period: Overall Study
Arm/Group | FMP1/AS02A Malaria Vaccine 10ug (Cohort A) | Imovax (Cohort A) | FMP1/AS02A Malaria Vaccine 25 ug (Cohort B) | Imovax (Cohort B) | FMP1/AS02A Malaria Vaccine 50 ug (Cohort C) | Imovax (Cohort C)
Started | 30 | 15 | 30 | 15 | 30 | 15
Completed | 26 | 12 | 27 | 13 | 22 | 12
Not Completed | 4 | 3 | 3 | 2 | 8 | 3
Not completed — Withdrawal by Subject | 2 | 1 | 2 | 1 | 3 | 1
Not completed — Relocation | 1 | 0 | 1 | 1 | 5 | 2
Not completed — Death | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 0 | 2 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: one subject from FMP1/AS02A Cohort A withdrew after randomization and prior to baseline measurement
Groups:
- Total: Total of all reporting groups
Arm/Group | FMP1/AS02A Malaria Vaccine 10ug (Cohort A) | Imovax (Cohort A) | FMP1/AS02A Malaria Vaccine 25 ug (Cohort B) | Imovax (Cohort B) | FMP1/AS02A Malaria Vaccine 50 ug (Cohort C) | Imovax (Cohort C) | Total
Number analyzed (Participants) | 29 | 15 | 30 | 15 | 30 | 15 | 134
Age, Continuous [Mean (Standard Deviation); unit: Months] | 28.5 (9.6) | 28.8 (9.7) | 29.5 (10.9) | 29.9 (11.2) | 29.0 (9.9) | 29.2 (10.9) | 29.0 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 8 | 19 | 9 | 13 | 10 | 76
  Male | 12 | 7 | 11 | 6 | 17 | 5 | 58
Region of Enrollment [Number; unit: participants]
  Kenya | 29 | 15 | 30 | 15 | 30 | 15 | 134
Temperature (celcius) [Mean (Standard Deviation); unit: Celcius] | 36.36 (0.42) | 36.30 (36.49) | 36.49 (0.57) | 36.46 (0.51) | 36.50 (0.62) | 36.85 (0.65) | 36.45 (0.54)
Pulse (bpm) [Mean (Standard Deviation); unit: beats per minute (bpm)] | 111.8 (21.4) | 102.7 (24.4) | 108.8 (14.1) | 116.5 (18.0) | 102.9 (17.3) | 119.7 (19.0) | 107.8 (18.0)
Respiratory rate (bpm) [Mean (Standard Deviation); unit: breaths per minute (bpm)] | 31.5 (5.3) | 30.9 (5.5) | 31.1 (5.3) | 29.9 (2.8) | 31.6 (5.2) | 32.8 (5.4) | 31.4 (5.2)
Systolic blood pressure (mmHg) [Mean (Standard Deviation); unit: mmHg] | 96.6 (9.2) | 96.4 (14.5) | 95.2 (9.6) | 96.1 (11.8) | 97.3 (11.7) | 94.4 (14.1) | 96.4 (10.1)
Diastolic blood pressure (mmHg) [Mean (Standard Deviation); unit: mmHg] | 55.8 (11.0) | 54.5 (11.5) | 51.3 (7.5) | 53.3 (10.1) | 53.5 (10.2) | 52.0 (8.0) | 53.5 (9.7)
Height (cm) [Mean (Standard Deviation); unit: cm] | 84.7 (7.0) | 84.3 (6.7) | 84.8 (9.0) | 85.7 (9.2) | 83.1 (6.9) | 81.2 (8.3) | 84.2 (7.6)
Weight (kg) [Mean (Standard Deviation); unit: kg] | 12.23 (1.97) | 11.97 (2.10) | 12.04 (2.52) | 12.51 (3.11) | 11.73 (1.93) | 11.04 (2.17) | 12.00 (2.14)

OUTCOME MEASURES:

1. Primary Outcome: Occurrence of Solicited Symptoms During a 8 Day Follow-up Period After Each Vaccination
Description: Occurrence of any, local, or general solicited symptoms during the 8 day follow-up period
Time Frame: 40 days
Measure: Number; unit: events
Groups:
- FMP1/AS02A Malaria Vaccine: Subject vaccinated with FMP1/AS02A (cohorts A, B, and C)
- Imovax Rabies Vaccine: Subject vaccinated with Imovax Rabies Vaccine (cohorts A, B, and C)
- Overall: Subjects vaccinated with FMP1/AS02A and Imovax Rabies Vaccine (cohorts A, B, and C)
Arm/Group | FMP1/AS02A Malaria Vaccine | Imovax Rabies Vaccine | Overall
Number analyzed (Participants) | 90 | 45 | 135
events
  Cohort A: Any Imm - Any Symptom | 24 | 11 | 35
  Cohort A: Any Imm - Local | 15 | 2 | 17
  Cohort A: Any Imm - General | 18 | 10 | 29
  Cohort A: Imm 1 - Any Symptom | 16 | 7 | 23
  Cohort A: Imm 1 - Local | 9 | 0 | 9
  Cohort A: Imm 1 - General | 11 | 7 | 18
  Cohort A: Imm 2 - Any Symptom | 13 | 6 | 19
  Cohort A: Imm 2 - Local | 5 | 2 | 7
  Cohort A: Imm 2 - General | 10 | 4 | 14
  Cohort A: Imm 3 - Any Symptom | 4 | 2 | 6
  Cohort A: Imm 3 - Local | 1 | 0 | 1
  Cohort A: Imm 3 - General | 4 | 2 | 6
  Cohort B: Any Imm - Any Symptom | 28 | 10 | 38
  Cohort B: Any Imm - Local | 24 | 1 | 25
  Cohort B: Any Imm - General | 18 | 10 | 28
  Cohort B: Imm 1 - Any Symptom | 21 | 6 | 27
  Cohort B: Imm 1 - Local | 14 | 0 | 14
  Cohort B: Imm 1 - General | 12 | 6 | 18
  Cohort B: Imm 2 - Any Symptom | 15 | 5 | 20
  Cohort B: Imm 2 - Local | 12 | 1 | 13
  Cohort B: Imm 2 - General | 8 | 5 | 13
  Cohort B: Imm 3 - Any Symptom | 15 | 4 | 19
  Cohort B: Imm 3 - Local | 11 | 0 | 11
  Cohort B: Imm 3 - General | 7 | 4 | 11
  Cohort C: Any Imm - Any Symptom | 28 | 8 | 36
  Cohort C: Any Imm - Local | 26 | 2 | 28
  Cohort C: Any Imm - General | 20 | 6 | 26
  Cohort C: Imm 1 - Any Symptom | 24 | 4 | 28
  Cohort C: Imm 1 - Local | 18 | 1 | 19
  Cohort C: Imm 1 - General | 15 | 3 | 18
  Cohort C: Imm 2 - Any Symptom | 19 | 4 | 23
  Cohort C: Imm 2 - Local | 17 | 1 | 18
  Cohort C: Imm 2 - General | 10 | 3 | 13
  Cohort C: Imm 3 - Any Symptom | 22 | 2 | 24
  Cohort C: Imm 3 - Local | 19 | 0 | 19
  Cohort C: Imm 3 - General | 10 | 2 | 12

2. Primary Outcome: Occurrence of Unsolicited Symptoms During a 30 Day Follow-up Period After Each Vaccination
Description: Occurrence of unsolicited symptoms during a 30 day follow-up period after each vaccination (day of vaccination and the 29 subsequent days)
Time Frame: 90 days
Measure: Number; unit: events
Groups:
- FMP1/AS02A Imm 1: Subjects 1st vaccination with FMP1/AS02A
- FMP1/AS02A Imm 2: Subjects 2nd vaccination with FMP1/AS02A
- FMP1/AS02A Imm 3: Subjects 3rd vaccination with FMP1/AS02A
- FMP1/AS02A Any Imm; Imovax Any Imm: Subjects vaccinated within all immunization cycles
- Imovax Imm 1: Subjects 1st vaccination with Imovax Rabies Vaccine
- Imovax Imm 2: Subjects 2nd vaccination with Imovax Rabies Vaccine
- Imovax Imm 3: Subjects 3rd vaccination with Imovax Rabies Vaccine
Arm/Group | FMP1/AS02A Imm 1 | FMP1/AS02A Imm 2 | FMP1/AS02A Imm 3 | FMP1/AS02A Any Imm | Imovax Imm 1 | Imovax Imm 2 | Imovax Imm 3 | Imovax Any Imm
Number analyzed (Participants) | 30 | 30 | 28 | 88 | 15 | 14 | 13 | 42
events
  Cohort A: Parasitic Infection | 19 | 15 | 13 | 27 | 9 | 5 | 8 | 13
  Cohort A: Resistance Mechanism | 13 | 18 | 14 | 28 | 5 | 7 | 4 | 10
  Cohort A: Skin and appendages | 7 | 14 | 11 | 20 | 8 | 5 | 4 | 11
  Cohort A: Respiratory System | 10 | 8 | 4 | 18 | 5 | 7 | 2 | 11
  Cohort A: Gastrointestinal System | 7 | 9 | 4 | 17 | 0 | 3 | 6 | 7
  Cohort A: Body as a Whole: General | 5 | 6 | 2 | 10 | 2 | 2 | 1 | 4
  Cohort A: Vision | 0 | 4 | 2 | 6 | 2 | 1 | 1 | 4
  Cohort A: Red Blood Cells | 1 | 1 | 2 | 4 | 0 | 0 | 0 | 0
  Cohort A: Unclassified | 0 | 1 | 1 | 2 | 1 | 0 | 0 | 1
  Cohort A: Application Site | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 1
  Cohort A: Urinary System | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 0
  Cohort B: Resistance Mechnism | 14 | 15 | 13 | 24 | 7 | 11 | 7 | 15
  Cohort B: Parasitic Infection | 14 | 14 | 12 | 25 | 9 | 7 | 6 | 13
  Cohort B: Skin and Appedages | 11 | 13 | 5 | 20 | 5 | 5 | 4 | 8
  Cohort B: Respiratory System | 11 | 13 | 5 | 20 | 5 | 5 | 4 | 8
  Cohort B: Gastrointestinal System | 6 | 6 | 5 | 13 | 2 | 1 | 3 | 6
  Cohort B: Body as a Whole: General | 8 | 4 | 3 | 12 | 1 | 1 | 3 | 4
  Cohort B: Vision | 1 | 7 | 4 | 11 | 2 | 2 | 1 | 5
  Cohort B: Liver and Biliary System | 1 | 0 | 3 | 4 | 1 | 1 | 0 | 2
  Cohort B: Unclassified | 1 | 0 | 2 | 3 | 2 | 0 | 1 | 3
  Cohort B: Musculoskeletal System | 1 | 1 | 1 | 3 | 0 | 0 | 0 | 0
  Cohort B: Red Blood Cells | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2
  Cohort B: Central and Peripheral Nervous | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1
  Cohort B: Hearing and Vestibular | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Cohort B: Urinary System | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Cohort C: Resistance Mechanism | 18 | 18 | 10 | 25 | 8 | 7 | 8 | 13
  Cohort C: Parasitic Infection | 14 | 11 | 8 | 17 | 10 | 10 | 7 | 13
  Cohort C: Skin and Appendages | 9 | 12 | 2 | 17 | 5 | 4 | 4 | 10
  Cohort C: Respiratory System | 10 | 1 | 4 | 12 | 7 | 3 | 3 | 10
  Cohort C: Gastrointestinal System | 2 | 8 | 5 | 12 | 3 | 2 | 5 | 8
  Cohort C: Body as a Whole: General | 4 | 4 | 3 | 10 | 1 | 1 | 2 | 3
  Cohort C: Vision | 7 | 1 | 1 | 8 | 2 | 2 | 0 | 4
  Cohort C: Unclassified | 1 | 2 | 3 | 6 | 1 | 0 | 1 | 2
  Cohort C: Hearing and Vestibular | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 1
  Cohort C: Red Blood Cells | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 1
  Cohort C: Central and Peripheral Nervous | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
  Cohort C: Liver and Biliary System | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
  Cohort C: Urinary System | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0

3. Primary Outcome: Occurrence of Serious Adverse Events During an 8 Month Follow-up Period Following the First Dose of Study Vaccine
Description: Occurrence of solicited and unsolicited serious adverse events during an 8 month follow-up period following the first dose of study vaccine
Time Frame: 8 months
Measure: Number; unit: events
Groups:
- FMP1/AS02A Malaria Vaccine: Subject vaccinated with FMP1/AS02A
- Imovax Rabies Vaccine: Subject vaccinated with Imovax Rabies Vaccine
- Overall: Subjects vaccinated with FMP1/AS02A and Imovax Rabies Vaccine
Arm/Group | FMP1/AS02A Malaria Vaccine | Imovax Rabies Vaccine | Overall
Number analyzed (Participants) | 89 | 45 | 134
events
  Cohort A: Any SAE | 2 | 1 | 3
  Cohort A: Imm 1 | 0 | 0 | 0
  Cohort A: Imm 2 | 1 | 0 | 1
  Cohort A: Imm 3 | 1 | 1 | 2
  Cohort B: Any SAE | 0 | 0 | 0
  Cohort B: Imm 1 | 0 | 0 | 0
  Cohort B: Imm 2 | 0 | 0 | 0
  Cohort B: Imm 3 | 0 | 0 | 0
  Cohort C: Any SAE | 1 | 0 | 1
  Cohort C: Imm 1 | 0 | 0 | 0
  Cohort C: Imm 2 | 1 | 0 | 1
  Cohort C: Imm 3 | 0 | 0 | 0

4. Secondary Outcome: Anti-FMP1 Antibody Titer Responses
Description: Antibody responses to FMP1 by ELISA following immunization with the study vaccine through 364 days following the first dose of study vaccine
Time Frame: 364 days
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | FMP1/AS02A Malaria Vaccine 10ug (Cohort A) | Imovax (Cohort A) | FMP1/AS02A Malaria Vaccine 25 ug (Cohort B) | Imovax (Cohort B) | FMP1/AS02A Malaria Vaccine 50 ug (Cohort C) | Imovax (Cohort C)
Number analyzed (Participants) | 29 | 15 | 30 | 15 | 30 | 15
titers
  Pre-Imm 1 | 2141 [1090 to 4205] | 2814 [827 to 9757] | 2737 [1492 to 5023] | 3226 [1250 to 8328] | 2301 [1074 to 4930] | 1041 [319 to 3401]
  Day 14 | 2711 [1524 to 4824] | 2857 [827 to 9757] | 4784 [2702 to 8469] | 2520 [835 to 7604] | 5729 [3320 to 9887] | 944 [361 to 2470]
  Pre-Imm 2 | 2440 [1449 to 41088] | 2829 [832 to 9611] | 2777 [1522 to 5065] | 4282 [1465 to 12516] | 4705 [2870 to 7714] | 1041 [396 to 2731]
  Day 44 | 4438 [2579 to 7637] | 2562 [724 to 9067] | 8390 [4733 to 14874] | 3593 [1185 to 10894] | 10791 [5421 to 21479] | 1105 [384 to 3178]
  Pre-Imm 3 | 4534 [2854 to 7202] | 2013 [412 to 9832] | 10240 [6409 to 16360] | 2258 [780 to 6537] | 10631 [5599 to 20184] | 1034 [388 to 2751]
  Day 74 | 10151 [6328 to 16285] | 1529 [421 to 5546] | 43399 [29132 to 64653] | 3368 [1295 to 8758] | 50166 [28307 to 88906] | 790 [306 to 2039]
  Day 90 | 10332 [5944 to 17960] | 1768 [431 to 7246] | 27189 [17827 to 41468] | 2909 [1251 to 8765] | 34657 [18914 to 63305] | 1039 [371 to 2910]
  Day 180 | 5354 [2954 to 9702] | 1788 [514 to 6213] | 13496 [8514 to 21392] | 4318 [1532 to 12170] | 14840 [7481 to 29434] | 999 [443 to 2257]
  Day 270 | 6190 [3520 to 10886] | 1877 [484 to 7278] | 14839 [8301 to 26527] | 6020 [2142 to 16921] | 15380 [8127 to 29108] | 1970 [659 to 5891]
  Day 364 | 4115 [2235 to 7574] | 2238 [641 to 7812] | 12043 [6585 to 22027] | 4005 [1351 to 11872] | 8807 [4083 to 18996] | 1295 [399 to 4204]

ADVERSE EVENTS:
Time Frame: 240 days
Description: The numbers of participants experiencing each specific event is not known, only the number of occurrences of each event. Therefore, individual occurrences are listed separately in the tables
Groups:
- Imovax: Subject vaccinated with Imovax Rabies Vaccine
Arm/Group | FMP1/AS02A Malaria Vaccine | Imovax
All-Cause Mortality (participants affected / at risk) | 1/90 | 0/45
Serious Adverse Events (participants affected / at risk) | 3/90 | 2/45
Other Adverse Events (participants affected / at risk) | 87/90 | 10/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FMP1/AS02A Malaria Vaccine (N=90) | Imovax (N=45)
Convulsions (Nervous system disorders) | 1 (1) | 0 (0) — Cohort A, Imm 3
Anemia (General disorders) | 1 (1) | 0 (0) — Cohort A, Imm 3 (death from Anemia)
Convulsions (Nervous system disorders) | 1 (1) | 0 (0) — Cohort A, Imm 2
Convulstions (Nervous system disorders) | 1 (1) | 0 (0) — Cohort C, Imm 2
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Cohort A, Imm 3
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) — Cohort A, Imm 3
Convulsions (Nervous system disorders) | 0 (0) | 1 (1) — Cohort B, Imm 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FMP1/AS02A Malaria Vaccine (N=90) | Imovax (N=45)
Fever (General disorders) | 1 (1) | 0 (0) — Cohort A, Imm 1
Loss of appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) — Cohort A, Imm 1
Pain at injection site (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Cohort A, Imm 1
Fever (General disorders) | 1 (1) | 0 (0) — Cohort A, Imm 2
Loss of appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) — Cohort A, Imm 2
Pain at injection site (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Cohort A, Imm 2
Swelling at injection site (General disorders) | 1 (1) | 0 (0) — Cohort A, Imm 2
Pain at the injection site (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Cohort A, Imm 3
Fever (General disorders) | 1 (1) | 0 (0) — Cohort A, Imm 3
Irritability (General disorders) | 1 (1) | 0 (0) — Cohort A, Imm 3
Loss of appetate (Metabolism and nutrition disorders) | 1 (1) | 0 (0) — Cohort A, Imm 3
Loss of appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) — Cohort A, Imm 3
Swelling at injection site (General disorders) | 1 (1) | 0 (0) — Cohort A, Imm 1
Pain at injections site (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Cohort A, Imm 2
Irritability (General disorders) | 1 (1) | 0 (0) — Cohort A, Imm 2
Fever (General disorders) | 1 (1) | 0 (0) — Cohort B, Imm 1
Pain at injection site (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Cohort B, Imm 2
Swelling at injection site (General disorders) | 1 (1) | 0 (0) — Cohort B, Imm 2
Loss of appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) — Cohort B, Imm 2
Loss of appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) — Cohort B, Imm 1
Pain at the injection site (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Cohort B, Imm 2
Pain at injection site (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Cohort B, Imm 3
Swelling at injection site (General disorders) | 1 (1) | 0 (0) — Cohort B, Imm 3
Loss of appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) — Cohort B, Imm 3
Pain at injection site (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Cohort B, Imm 1
Swelling at injection site (General disorders) | 1 (1) | 0 (0) — Cohort B, Imm 1
Irritability (General disorders) | 1 (1) | 0 (0) — Cohort B, Imm 1
Fever (General disorders) | 1 (1) | 0 (0) — Cohort B, Imm 2
Fever (General disorders) | 1 (1) | 0 (0) — Cohort B, Imm 3
Irritability (General disorders) | 1 (1) | 0 (0) — Cohort B, Imm 2
Pain at injection site (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Cohort C, Imm 1
Swelling at injection site (General disorders) | 1 (1) | 0 (0) — Cohort C, Imm 1
Fever (General disorders) | 1 (1) | 0 (0) — Cohort C, Imm 1
Pain at injection site (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Cohort C, Imm 2
Pain at injection site (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Cohort C, Imm 3
Fever (General disorders) | 1 (1) | 0 (0) — Cohort C, Imm 3
Pain at injection site (Infections and infestations) | 1 (1) | 0 (0) — Cohort C, Imm 1
Loss of appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) — Cohort C, Imm 2
Swelling at injection site (General disorders) | 1 (1) | 0 (0) — Cohort C, Imm 3
Loss of appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) — Cohort C, Imm 1
Fever (General disorders) | 1 (1) | 0 (0) — Cohort C, Imm 2
Swelling at injection site (General disorders) | 1 (1) | 0 (0) — Cohort C, Imm 2
Loss of appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) — Cohort C, Imm 3
Irritability (General disorders) | 1 (1) | 0 (0) — Cohort C, Imm 3
Pain at the injection site (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Cohort C, Imm 3
Pain at the injection site (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Cohort C, Imm 2
Swelling at injection site (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Cohort C, Imm 3
Loss of appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) — Cohort A, Imm 1
Fever (General disorders) | 0 (0) | 1 (1) — Cohort A, Imm 3
Fever (General disorders) | 0 (0) | 1 (1) — Cohort A, Imm 2
Fever (General disorders) | 0 (0) | 1 (1) — Cohort A, Imm 1
Loss of appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) — Cohort A, Imm 2
Pain at injection site (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Cohort A, Imm 2
Loss of appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) — Cohort B, Imm 2
Fever (General disorders) | 0 (0) | 1 (1) — Cohort B, Imm 3
Fever (General disorders) | 0 (0) | 1 (1) — Cohort B, Imm 1
Loss of appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) — Cohort B, Imm 1
Loss of appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) — Cohort A, Imm 3
Irritability (General disorders) | 0 (0) | 1 (1) — Cohort B, Imm 2
Loss of appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) — Cohort B, Imm 3
Fever (General disorders) | 0 (0) | 1 (1) — Cohort B, Imm 2
Pain at injection site (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Cohort B, Imm 2
Loss of appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) — Cohort C, Imm 2
Pain at injection site (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Cohort C, Imm 2
Fever (General disorders) | 0 (0) | 1 (1) — Cohort C, Imm 1
Fever (General disorders) | 0 (0) | 1 (1) — Cohort C, Imm 3
Loss of appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) — Cohort C, Imm 3
Fever (General disorders) | 0 (0) | 1 (1) — Cohort C, Imm 2
Pain at injection site (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Cohort C, Imm 1
Malaria (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — Cohort A, Imm 1
Rash pustular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Cohort A, Imm 2
Malaria (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — Cohort A, Imm 2
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — Cohort A, Imm 3
Coughing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Cohort A, Imm 1
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Cohort A, Imm 1
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Cohort A, Imm 1
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) — Cohort A, Imm 2
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Cohort A, Imm 2
Fever (General disorders) | 1 (1) | 0 (0) — Cohort A, Imm 2
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Cohort A, Imm 1
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — Cohort A, Imm 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Cohort A, Imm 2
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Cohort A, Imm 3
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Cohort A, Imm 3
Fever (General disorders) | 1 (1) | 0 (0) — Cohort A, Imm 1
Loss of appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) — Cohort A, Imm 2
Gingivitis (Gastrointestinal disorders) | 1 (1) | 0 (0) — Cohort A, Imm 2
Oral candidiasis (Gastrointestinal disorders) | 1 (1) | 0 (0) — Cohort A, Imm 2
Upper respiratory tract infection (Gastrointestinal disorders) | 1 (1) | 0 (0) — Cohort A, Imm 3
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) — Cohort A, Imm 1
Superficial burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Cohort A, Imm 3
Folliculitis (Infections and infestations) | 1 (1) | 0 (0) — Cohort A, Imm 3
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) — Cohort A, Imm 3
Poor feeding (General disorders) | 1 (1) | 0 (0) — Cohort A, Imm 3
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0) — Cohort A, Imm 2
Small plaques (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Cohort A, Imm 2
Malaria (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — Cohort A, Imm 3
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0) — Cohort A, Imm 1
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Cohort A, Imm 2
Coughing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Cohort A, Imm 3
Furunculosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Cohort A, Imm 1
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) — Cohort A, Imm 1
Injection site induration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Cohort A, Imm 2
Micturition disorder (Renal and urinary disorders) | 1 (1) | 0 (0) — Cohort A, Imm 2
Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Cohort A, Imm 3
Rash pustular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Cohort A, Imm 3
Otitis media (Infections and infestations) | 1 (1) | 0 (0) — Cohort A, Imm 2
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Cohort A, Imm 3
Gastroenteritis (Gastrointestinal disorders) | 1 (1) | 0 (0) — Cohort A, Imm 3
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Cohort A, Imm 3
Loss of appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) — Cohort A, Imm 1
Folliculitis (Infections and infestations) | 1 (1) | 0 (0) — Cohort A, Imm 2
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) — Cohort A, Imm 2
Loss of appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) — Cohort A, Imm 3
Coughing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Cohort A, Imm 2
Otitis externa (Ear and labyrinth disorders) | 1 (1) | 0 (0) — Cohort A, Imm 1
Laryngitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Cohort A, Imm 2
Folliculitis (Infections and infestations) | 1 (1) | 0 (0) — Cohort A, Imm 1
Foriegn body in throat (Gastrointestinal disorders) | 1 (1) | 0 (0) — Cohort A, Imm 2
Enterobiasis (Gastrointestinal disorders) | 1 (1) | 0 (0) — Cohort A, Imm 3
Otitis media (Infections and infestations) | 1 (1) | 0 (0) — Cohort A, Imm 3
Rash pustular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Cohort A, Imm 1
Tinea corporis (Infections and infestations) | 1 (1) | 0 (0) — Cohort A, Imm 3
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Cohort A, Imm 1
Stomatitis ulcerative (Gastrointestinal disorders) | 1 (1) | 0 (0) — Cohort A, Imm 2
Moniliasis (Infections and infestations) | 1 (1) | 0 (0) — Cohort A, Imm 1
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0) — Cohort A, Imm 3
Fever (General disorders) | 1 (1) | 0 (0) — Cohort A, Imm 3
Moniliasis (Infections and infestations) | 1 (1) | 0 (0) — Cohort A, Imm 3
Gastroenteritis (Gastrointestinal disorders) | 1 (1) | 0 (0) — Cohort A, Post-1
Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Cohort A, Imm 1
Marlaria (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — Cohort A, Imm 2
Eye pain (Eye disorders) | 1 (1) | 0 (0) — Cohort A, Imm 2
Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Cohort A, Imm 2
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) — Cohort A, Imm 1
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) — Cohort A, Imm 1
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) — Cohort A, Imm 1
Infection (Infections and infestations) | 1 (1) | 0 (0) — Cohort A, Imm 2
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — Cohort A, Imm 2
Urinary tract infection (Renal and urinary disorders) | 1 (1) | 0 (0) — Cohort A, Imm 3
Urinary tract infection (Renal and urinary disorders) | 1 (1) | 0 (0) — Cohort A, Imm 1
Foriegn body in nostril (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Cohort A, Imm 1
Tinea corporis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Cohort A, Imm 1
Pain (General disorders) | 1 (1) | 0 (0) — Cohort A, Imm 1
Herpes simplex (Infections and infestations) | 1 (1) | 0 (0) — Cohort A, Imm 2
Conjunctivtis (Infections and infestations) | 1 (1) | 0 (0) — Cohort A, Imm 3
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Cohort B, Imm 1
Folliculitis (Infections and infestations) | 1 (1) | 0 (0) — Cohort B, Imm 1
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Cohort B, Imm 2
Malaria (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — Cohort B, Imm 2
Tinea corporis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Cohort B, Imm 2
History of fever (General disorders) | 1 (1) | 0 (0) — Cohort B, Imm 3
Malaria (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — Cohort B, Imm 3
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Cohort B, Imm 3
History of fever (General disorders) | 1 (1) | 0 (0) — Cohort B, Imm 2
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Cohort B, Imm 1
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Cohort B, Imm 1
Loose stool (Gastrointestinal disorders) | 1 (1) | 0 (0) — Cohort B, Imm 2
Folliculitis (Infections and infestations) | 1 (1) | 0 (0) — Cohort B, Imm 2
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Cohort B, Imm 2
Moniliasis (Infections and infestations) | 1 (1) | 0 (0) — Cohort B, Post-1
Poor feeding (General disorders) | 1 (1) | 0 (0) — Cohort B, Imm 1
Coughing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Cohort B, Pre-1
Loss of appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) — Cohort B, Imm 1
Rash pustular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Cohort B, Imm 1
Gastroenteritis (Gastrointestinal disorders) | 1 (1) | 0 (0) — Cohort B, Imm 2
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) — Cohort B, Imm 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Cohort B, Imm 3
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) — Cohort B, Imm 1
Malaria (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — Cohort B, Imm 1
Loss of appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) — Cohort B, Imm 2
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) — Cohort B, Imm 2
Loss of appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) — Cohort B, Imm 3
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0) — Cohort B, Imm 3
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0) — Cohort B, Imm 2
Gastroenteritis (Gastrointestinal disorders) | 1 (1) | 0 (0) — Cohort B, Imm 3
Rash pustular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Cohort B, Pre-1
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) — Cohort B, Imm 1
Coughing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Cohort B, Imm 1
Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Cohort B, Imm 1
Moniliasis (Infections and infestations) | 1 (1) | 0 (0) — Cohort B, Imm 2
Otitis externa (Ear and labyrinth disorders) | 1 (1) | 0 (0) — Cohort B, Imm 2
Folliculitis (Infections and infestations) | 1 (1) | 0 (0) — Cohort B, Post-1
Coughing (Reproductive system and breast disorders) | 1 (1) | 0 (0) — Cohort B, Imm 1
History of fever (General disorders) | 1 (1) | 0 (0) — Cohort B, Imm 1
Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Cohort B, Imm 3
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Cohort B, Imm 1
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0) — Cohort B, Imm 1
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Cohort B, Imm 3
SBPT increased (Investigations) | 1 (1) | 0 (0) — Cohort B, Imm 3
Rash pustular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Cohort B, Imm 3
Septic lesion left pinna (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Cohort B, Imm 1
Rash pustular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Cohort B, Imm 2
Tinea capitis (Infections and infestations) | 1 (1) | 0 (0) — Cohort B, Imm 2
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) — Cohort B, Imm 3
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) — Cohort B, Imm 1
Helminthiasis (Infections and infestations) | 1 (1) | 0 (0) — Cohort B, Imm 2
Stomatitis ulceratived (Gastrointestinal disorders) | 1 (1) | 0 (0) — Cohort B, Imm 2
Micturition disorder (Renal and urinary disorders) | 1 (1) | 0 (0) — Cohort B, Imm 3
Folliculitis (Infections and infestations) | 1 (1) | 0 (0) — Cohort B, Imm 3
Helminthiasis (Infections and infestations) | 1 (1) | 0 (0) — Cohort B, Imm 3
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Cohort B, Pre-1
Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Cohort B, Imm 2
Tinea corporis (Infections and infestations) | 1 (1) | 0 (0) — Cohort B, Imm 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Cohort B, Imm 2
Rectal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0) — Cohort B, Pre-1
SGPT increased (Investigations) | 1 (1) | 0 (0) — Cohort B, Imm 3
Poor feeding (General disorders) | 1 (1) | 0 (0) — Cohort B, Imm 3
Conjuctivitis (Infections and infestations) | 1 (1) | 0 (0) — Cohort B, Imm 2
Loss of appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) — Cohort B, Post-1
Rash pustular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Cohort B, Post-1
SGPT increased (Investigations) | 1 (1) | 0 (0) — Cohort B, Imm 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Cohort B, Imm 1
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Cohort B, Post-1
Coughing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Cohort B, Imm 2
Otitis media (Infections and infestations) | 1 (1) | 0 (0) — Cohort B, Imm 3
Otitis media (Infections and infestations) | 1 (1) | 0 (0) — Cohort B, Imm 2
Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Cohort C, Imm 1
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Cohort C, Imm 1
Rash pustular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Cohort C, Imm 1
Malaria (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — Cohort C, Imm 2
Rash pustular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Cohort C, Imm 2
Poor feeding (General disorders) | 1 (1) | 0 (0) — Cohort C, Imm 2
Folliculitis (Infections and infestations) | 1 (1) | 0 (0) — Cohort C, Imm 2
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Cohort C, Imm 2
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Cohort C, Imm 3
Malaria (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — Cohort C, Imm 1
Abscess (Infections and infestations) | 1 (1) | 0 (0) — Cohort C, Imm 2
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — Cohort C, Imm 2
Loss of appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) — Cohort C, Imm 2
Gluteal ulcer (General disorders) | 1 (1) | 0 (0) — Cohort C, Imm 3
Gastroenteritis (Gastrointestinal disorders) | 1 (1) | 0 (0) — Cohort C, Imm 3
Malaria (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — Cohort C, Imm 3
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Cohort C, Imm 1
Loose stool (Gastrointestinal disorders) | 1 (1) | 0 (0) — Cohort C, Imm 3
Poor feeding (General disorders) | 1 (1) | 0 (0) — Cohort C, Imm 3
Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Cohort C, Imm 3
Gastroenteritis (Gastrointestinal disorders) | 1 (1) | 0 (0) — Cohort C, Imm 1
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) — Cohort C, Imm 2
Herpes simplex (Infections and infestations) | 1 (1) | 0 (0) — Cohort C, Imm 2
History of fever (General disorders) | 1 (1) | 0 (0) — Cohort C, Imm 2
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Cohort C, Imm 3
Lower respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Cohort C, Imm 1
Helminthiasis (Infections and infestations) | 1 (1) | 0 (0) — Cohort C, Imm 2
Fever (General disorders) | 1 (1) | 0 (0) — Cohort C, Imm 2
Urinary tract infection (Renal and urinary disorders) | 1 (1) | 0 (0) — Cohort C, Imm 3
Coughing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Cohort C, Imm 1
Fever (General disorders) | 1 (1) | 0 (0) — Cohort C, Imm 1
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0) — Cohort C, Imm 3
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0) — Cohort C, Imm 1
Tinea corporis (Infections and infestations) | 1 (1) | 0 (0) — Cohort C, Imm 2
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) — Cohort C, Imm 2
Earache (Ear and labyrinth disorders) | 1 (1) | 0 (0) — Cohort C, Imm 2
Upper resporatory tract infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Cohort C, Imm 3
Loss of appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) — Cohort C, Imm 1
Tinea capitis (Infections and infestations) | 1 (1) | 0 (0) — Cohort C, Imm 2
Folliculitis (Infections and infestations) | 1 (1) | 0 (0) — Cohort C, Imm 3
Otitis media (Infections and infestations) | 1 (1) | 0 (0) — Cohort C, Imm 1
Marlaria (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — Cohort C, Imm 1
History of fever (Gastrointestinal disorders) | 1 (1) | 0 (0) — Cohort C, Imm 3
Upper respriatory tract infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Cohort C, Imm 2
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0) — Cohort C, Imm 2
Loss of appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) — Cohort C, Imm 3
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) — Cohort C, Imm 3
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) — Cohort C, Imm 2
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Cohort C, Imm 2
Headache (Nervous system disorders) | 1 (1) | 0 (0) — Cohort C, Imm 2
Rash pustular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Cohort C, Imm 3
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) — Cohort C, Imm 3
Coughing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Cohort C, Imm 2
Coughing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Cohort C, Imm 3
Tinea capitis (Infections and infestations) | 1 (1) | 0 (0) — Cohort C, Imm 1
Conjunctivitis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Cohort C, Imm 1
Septic wound secondary to trauma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Cohort C, Imm 2
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) — Cohort C, Imm 2
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) — Cohort C, Imm 2
Folliculitis (Infections and infestations) | 1 (1) | 0 (0) — Cohort C, Imm 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Cohort A, Imm 1
Malaria (Blood and lymphatic system disorders) | 0 (0) | 1 (1) — Cohort A, Imm 1
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Cohort A, Imm 1
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Cohort A, Imm 2
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Cohort A, Imm 2
Malaria (Blood and lymphatic system disorders) | 0 (0) | 1 (1) — Cohort A, Imm 2
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) — Cohort A, Imm 2
Tinea corporis (Infections and infestations) | 0 (0) | 1 (1) — Cohort A, Imm 2
Malaria (Blood and lymphatic system disorders) | 0 (0) | 1 (1) — Cohort A, Imm 3
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Cohort A, Imm 1
Rash pustular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Cohort A, Imm 1
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1) — Cohort A, Imm 1
Gastroenteritis (Gastrointestinal disorders) | 0 (0) | 1 (1) — Cohort A, Imm 3
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) — Cohort A, Imm 1
Coughing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Cohort A, Imm 2
Rash pustular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Cohort A, Imm 2
Loss of appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) — Cohort A, Imm 3
Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Cohort A, Imm 1
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) — Cohort A, Imm 2
Upper respitratory tract infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Cohort A, Imm 2
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Cohort A, Imm 3
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) — Cohort A, Imm 3
Rash pustular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Cohort A, Imm 3
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Cohort A, Imm 1
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1) — Cohort A, Imm 2
Loss of appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) — Cohort A, Imm 2
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Cohort A, Imm 3
Helminthiasis (Infections and infestations) | 0 (0) | 1 (1) — Cohort A, Imm 1
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) — Cohort A, Imm 1
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) — Cohort A, Imm 2
Coughing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Cohort A, Imm 1
History of fever (General disorders) | 0 (0) | 1 (1) — Cohort A, Imm 3
Otitis externa (Ear and labyrinth disorders) | 0 (0) | 1 (1) — Cohort A, Imm 1
Anal fissure (Gastrointestinal disorders) | 0 (0) | 1 (1) — Cohort A, Imm 1
Pruritus (Gastrointestinal disorders) | 0 (0) | 1 (1) — Cohort A, Imm 1
Tinea capitis (Infections and infestations) | 0 (0) | 1 (1) — Cohort A, Imm 2
Superficial burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Cohort A, Imm 3
Injection site hyperpigmentation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Cohort A, Imm 1
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Cohort A, Imm 2
Coughing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Cohort A, Imm 3
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1) — Cohort A, Imm 3
Malaria (Blood and lymphatic system disorders) | 0 (0) | 1 (1) — Cohort B, Imm 1
Coughing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Cohort B, Imm 2
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Cohort B, Imm 2
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Cohort B, Imm 3
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Cohort B, Imm 3
Stomatitis ulcerative (Gastrointestinal disorders) | 0 (0) | 1 (1) — Cohort B, Imm 3
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1) — Cohort B, Imm 1
Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Cohort B, Imm 1
Coughing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Cohort B, Imm 1
Malaria (Blood and lymphatic system disorders) | 0 (0) | 1 (1) — Cohort B, Imm 2
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Cohort B, Imm 2
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1) — Cohort B, Imm 3
Rash pustular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Cohort B, Imm 3
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Cohort B, Imm 1
Poor feeding (General disorders) | 0 (0) | 1 (1) — Cohort B, Imm 1
Upper respitratory tract infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Cohort B, Imm 2
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1) — Cohort B, Imm 2
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) — Cohort B, Imm 2
Conjuntivitis (Infections and infestations) | 0 (0) | 1 (1) — Cohort B, Post-1
Hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1) — Cohort B, Imm 1
SGPT increased (Investigations) | 0 (0) | 1 (1) — Cohort B, Imm 1
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Cohort B, Post-1
Malaria (Blood and lymphatic system disorders) | 0 (0) | 1 (1) — Cohort B, Imm 3
Fever (General disorders) | 0 (0) | 1 (1) — Cohort B, Imm 3
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) — Cohort B, Imm 3
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) — Cohort B, Imm 2
Folliculitis (Infections and infestations) | 0 (0) | 1 (1) — Cohort B, Post-1
Rash pustular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Cohort B, Imm 1
Headache (Nervous system disorders) | 0 (0) | 1 (1) — Cohort B, Imm 1
Fever (General disorders) | 0 (0) | 1 (1) — Cohort B, Imm 2
Headache (Nervous system disorders) | 0 (0) | 1 (1) — Cohort B, Imm 2
Poor feeding (General disorders) | 0 (0) | 1 (1) — Cohort B, Imm 3
Folliculitis (Infections and infestations) | 0 (0) | 1 (1) — Cohort B, Imm 1
Folliculitis (Infections and infestations) | 0 (0) | 1 (1) — Cohort B, Imm 2
Coughing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Cohort B, Imm 3
Loose stool (Gastrointestinal disorders) | 0 (0) | 1 (1) — Cohort B, Imm 3
Pruritis ani (Infections and infestations) | 0 (0) | 1 (1) — Cohort B, Imm 3
Folliculitis (Infections and infestations) | 0 (0) | 1 (1) — Cohort B, Imm 3
Gastroenteritis (Gastrointestinal disorders) | 0 (0) | 1 (1) — Cohort B, Imm 3
Gingivitis (Infections and infestations) | 0 (0) | 1 (1) — Cohort B, Imm 1
Rhinitis (Infections and infestations) | 0 (0) | 1 (1) — Cohort B, Imm 1
Tinea capitis (Infections and infestations) | 0 (0) | 1 (1) — Cohort B, Imm 1
Rash pustular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Cohort B, Imm 2
Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Cohort B, Imm 3
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Cohort B, Imm 1
Tinea corporis (Infections and infestations) | 0 (0) | 1 (1) — Cohort B, Imm 2
SGPT increased (Investigations) | 0 (0) | 1 (1) — Cohort B, Imm 2
Urinary tract infection (Renal and urinary disorders) | 0 (0) | 1 (1) — Cohort B, Imm 2
Coryza (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Cohort C, Imm 1
Malaria (Blood and lymphatic system disorders) | 0 (0) | 1 (1) — Cohort C, Imm 1
Rash pustular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Cohort C, Imm 1
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Cohort C, Imm 1
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1) — Cohort C, Imm 2
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Cohort C, Imm 2
Coughing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Cohort C, Imm 2
History of fever (General disorders) | 0 (0) | 1 (1) — Cohort C, Imm 3
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) — Cohort C, Imm 3
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Cohort C, Imm 3
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Cohort C, Imm 1
Skin disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Cohort C, Imm 1
Malaria (Blood and lymphatic system disorders) | 0 (0) | 1 (1) — Cohort C, Imm 2
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) — Cohort C, Imm 2
Malaria (Blood and lymphatic system disorders) | 0 (0) | 1 (1) — Cohort C, Imm 3
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) — Cohort C, Imm 3
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Cohort C, Imm 3
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) — Cohort C, Imm 1
Rash pustular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Cohort C, Imm 2
Folliculitis (Infections and infestations) | 0 (0) | 1 (1) — Cohort C, Imm 3
Upper respriatory tract infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Cohort C, Imm 3
Coughing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Cohort C, Imm 1
Folliculitis (Infections and infestations) | 0 (0) | 1 (1) — Cohort C, Imm 1
Otitis exrterna (Ear and labyrinth disorders) | 0 (0) | 1 (1) — Cohort C, Imm 2
Gastroenteritis (Gastrointestinal disorders) | 0 (0) | 1 (1) — Cohort C, Imm 3
Poor feeding (General disorders) | 0 (0) | 1 (1) — Cohort C, Imm 3
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1) — Cohort C, Imm 1
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) — Cohort C, Imm 1
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Cohort C, Imm 2
Otitis externa (Ear and labyrinth disorders) | 0 (0) | 1 (1) — Cohort C, Imm 2
Folliculitis (Infections and infestations) | 0 (0) | 1 (1) — Cohort C, Imm 2
Fever (General disorders) | 0 (0) | 1 (1) — Cohort C, Imm 1
History of fever (General disorders) | 0 (0) | 1 (1) — Cohort C, Imm 2
tinea corporis (Infections and infestations) | 0 (0) | 1 (1) — Cohort C, Imm 2
Earache (Ear and labyrinth disorders) | 0 (0) | 1 (1) — Cohort C, Imm 3
Poor feeding (General disorders) | 0 (0) | 1 (1) — Cohort C, Imm 1
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) — Cohort C, Imm 1
Monilliasis (Infections and infestations) | 0 (0) | 1 (1) — Cohort C, Imm 2
Laryngitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Cohort C, Imm 1
Septic wound (Infections and infestations) | 0 (0) | 1 (1) — Cohort C, Imm 1
Helminthiasis (Infections and infestations) | 0 (0) | 1 (1) — Cohort C, Imm 2
Loss of appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) — Cohort C, Imm 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Cohort C, Imm 2
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) — Cohort C, Imm 3
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Cohort C, Imm 3
Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Cohort C, Imm 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No